CLINICAL TRIAL: NCT00157144
Title: Australia and New Zealand Adult Extracorporeal Membrane Oxygenation (ECMO) Audit 2005
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 186/04
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Distress Syndrome, Adult; Respiratory Insufficiency; Shock, Cardiogenic
Keywords: Lung Transplantation; Heart Transplantation
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Shock, Cardiogenic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is a means of artificially performing the function of the human lung and/or heart outside the body. Its use is escalating in a wide range of clinical settings in the adult population without evidence or guidelines to support this practice.

This study involves a nationwide questionnaire which has two components. The initial pilot survey will attempt to identify all institutions currently practicing ECMO or those intending to do so in the future, and are willing to participate in prospective data collection. The second phase will involve a monthly survey of these centres regarding the extent of ECMO use, practice details implemented, and outcome data.

It is hoped that the collection of this information will later assist in the development of guidelines for this expensive and presently unsubstantiated practice, together with the construction of appropriate training programs for staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ECMO in Australia and New Zealand

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent A Pellegrino, MBBS, Principal Investigator — National Health and Medical Research Council, Australia
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Hastings SL, Pellegrino VA, Preovolos A, Salamonsen RF. Survey of adult extracorporeal membrane oxygenation (ECMO) practice and attitudes among Australian and New Zealand intensivists. Crit Care Resusc. 2008 Mar;10(1):46. PMID 18304017